CLINICAL TRIAL: NCT02464956
Title: Feasibility of Production of Induced Pluripotent Stem Cell Derived Retinal Pigment Epithelial Cells Fulfilling Regulatory Requirements for Human Transplantation in Dry Age-related Macular Degeneration
Brief Title: Production of iPSC Derived RPE Cells for Transplantation in AMD
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: DACL1011
Record Dates: First submitted 2015-05-14; First posted 2015-06-08 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2021-09

CONDITIONS: Age Related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample and a skin sample will be collected from the study participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
No treatments exist for Age-related Macular Degeneration (AMD) when there is cell loss such as in late wet AMD or dry AMD. The differentiation of RPE cells from patient derived iPSC will offer valuable source of tissue for transplantation in these forms of AMD and may form basis for a future treatment option in terms of cell transplantation.

DETAILED DESCRIPTION:
It has been shown that adult human skin cells or human blood cells can be reprogrammed to become stem cells. This type of stem cell is called an induced Pluripotent Stem Cell (iPSC).It has been shown specifically that this type of stem cell can be produced from adult human skin cells or blood cells can in turn be converted into Retinal Pigment Epithelial (RPE) cells. These RPE cells are a very important cell type in the human retina that are abnormal and ultimately lost in Age-related Macular Degeneration (AMD). Although it has been shown to be possible to make RPE cells from adult human skin, it has not been done to a level to fulfil regulatory requirements for human transplantation in AMD.

This is a feasibility study involving 10 patients. The efficiency of creating an iPSC-Derived RPE cells from a patient's own skin or blood will be examined. A sample size of 10 patients will allow us to potentially consolidate the safety and efficacy of this method in order to create these cells within the context of a future transplantation trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 years
* Subjects with the ability to give informed consent
* Subjects with known AMD (both wet and dry)

Exclusion Criteria:

* Unable to give informed consent
* Subjects unable to give blood sample for medical reasons
* Subjects with coagulopathies
* Subjects who are known to be at risk of keloid scarring

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Age Related Macular Degeneration (AMD)
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Successful production of a Retinal Epithelial (RPE) layer that fulfils Regulatory Regulation for transplantation. This will be confirmed with standard laboratory characterisation of RPE and completed toxicity and safety studies on the cell layer. | 1 year